CLINICAL TRIAL: NCT01283295
Title: Immune Monitoring and Assay Development in Organ Transplant Recipients
Acronym: IMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Aneesh K. Mehta, Professor, Emory University
Other Study IDs: IRB00006248
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Organ Transplantation; Transplantation Immunology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs, serum, urine, kidney and liver biopsy samples, broncheolar lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Immune complications: Transplant recipients who develop a clinically recognized complication with potential immune etiology or ramifications. Examples include opportunistic infection, rejection, malignancy, alloantibody formation or immunosuppressive drug toxicity.
- Stable Transplant Recipient: Patients who demonstrate immune stability characterized by stable graft function without evident complication. These patients serve as comparators for Group 1
- Pre-Transplant Longitudinal: Patients who are candidates for kidney, pancreas, liver or lung transplant will be enrolled and followed longitudinally.
- Organ Donors: Donors for individuals meeting the criteria for Cohorts 1-3
- Disease state: Individuals with liver, renal or pulmonary diseases that may lead to the development or organ failure.
- Normal Volunteers

SUMMARY:
The purpose of this study to develop a well-characterized library of blood, biopsy tissue, and urine samples from transplant patients. Subjects without transplants will also be enrolled for comparison. Samples will be used to study the characteristics of patients undergoing transplantation that influence their response to transplant therapies and their reactions to drugs used in transplantation. This knowledge is important as it helps physicians design new drugs and tailor transplant therapies to the individual thereby reducing the side effects. In this study, people will be asked to donate blood, biopsy tissue and urine. Donation of these samples will not influence patients' treatments. These samples will be tested using a variety of biological tests to better understand how immunosuppressive drugs change the various components of the immune system. The tests will be for research only; no changes in an individual's treatment will be based on the results of tests performed in this study. If there is extra sample, the sample will be stored for use in other testing at a later date. The ultimate goal is find the right combination of medications for each individual patient while keeping their new organ working well. This study is a first step in that direction by perfecting tests used to characterize a patient's immune system

ELIGIBILITY:
Inclusion Criteria:

* Recipients of or candidates for organ transplantation or organ donors for recipients under evaluation at Emory University or CHOA
* Normal volunteers to include individuals without any known end-stage organ disease who are not on any immunosuppressive medication, and individuals with conditions requiring immunosuppression (i.e. dermatological diseases) that do not require transplant therapies
* Ability to understand the purposes and risks of the study and willingly give written informed consent, or in the case of minors, ability to give minor assent (children older than 5 years of age), in conjunction with written guardian consent

Exclusion Criteria:

* Patients who fail to meet the criteria for transplantation or post-transplant follow-up by Emory or Children's Healthcare of Atlanta physicians
* Any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating. Specific conditions include but are not limited to anemia prohibitive of phlebotomy, coagulopathy or technical considerations that would prevent acquisition of sufficient tissue on biopsy for clinical use, or medical urgency preventing timely administration of the consenting process.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric or adult organ transplant recipients, candidates for organ transplant, donors and normal volunteers of Emory University Hospital, the Emory Transplant Center or Children's Healthcare of Atlanta (CHOA)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To generate a bank of well-characterized biological samples from human subjects prior to or following organ transplantation for the purpose of subsequent evaluation using new and existing immunological assays | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh K Mehta, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No